CLINICAL TRIAL: NCT02321527
Title: Feasibility of Ultrasound Microbubble Contrast-Enhanced (CEUS) Ultrasound Sentinel Lymph Node Imaging With Guided Biopsy in Breast Cancer Patients
Brief Title: Feasibility of Ultrasound Microbubble Contrast-Enhanced (CEUS) Sentinel Lymph Node Imaging With Guided Biopsy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-0611; NCI-2015-00066 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Microbubble contrast-enhanced ultrasound; CEUS; Sentinel lymph nodes; SLN; Perflutren Protein-Type A Microspheres Injectable Suspension; OPTISON™; Ultrasound; Breast biopsy; Radioactive seed; Phone call; Fine needle aspiration; FNA
MeSH Terms: conditions — Breast Neoplasms | interventions — FS 069; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perflutren Protein-Type A Microspheres Injectable Suspension (Experimental): Participants receive a subdermal periareolar injection of 0.2 - 0.5 cc of microbubble contrast Perflutren Protein-Type A Microspheres Injectable Suspension (OPTISON™). Ultrasound images and videos of tumor and lymph nodes in underarm area taken. Biopsy of sentinel lymph node that was identified in ultrasound performed, and a titanium clip marker inserted into the node. After biopsy, a radioactive seed may be inserted into the node to allow surgeon to find and remove it during surgery. Participant called by phone 30 days after seed is removed to check for any side effects. This phone call should take about 10 minutes.
  Interventions: Drug: Perflutren Protein-Type A Microspheres Injectable Suspension; Device: Contrast-Enhanced Ultrasound (CEUS); Procedure: Biopsy + Radioactive Seed Placement; Behavioral: Phone Call

INTERVENTIONS:
Drug: Perflutren Protein-Type A Microspheres Injectable Suspension — Participants receive a subdermal periareolar injection of 0.2 - 0.5 cc of microbubble contrast Perflutren Protein-Type A Microspheres Injectable Suspension (OPTISON™) before breast ultrasound.
  Other Names: OPTISON
Device: Contrast-Enhanced Ultrasound (CEUS) — Ultrasound images of breast and videos of tumor and lymph nodes in underarm area taken after Perflutren Protein-Type A Microspheres Injectable Suspension injection.
Procedure: Biopsy + Radioactive Seed Placement — Biopsy of sentinel lymph node that was identified in ultrasound performed, and a titanium clip marker inserted into the node. After biopsy, a radioactive seed may be inserted into the node to allow surgeon to find and remove it during surgery.
Behavioral: Phone Call — Participant called by phone 30 days after seed is removed to check for any side effects. This phone call should take about 10 minutes.

SUMMARY:
The goal of this clinical research is to learn if an ultrasound contrast agent called OPTISON (perflutren protein type A) is effective in finding sentinel lymph nodes before surgery. Contrast agents can help make ultrasound images more accurate. The sentinel lymph node is the first node that may be the target of cancer cells that spread from the tumor.

DETAILED DESCRIPTION:
Study Procedures:

If you agree and are eligible to take part, you will receive perflutren protein type A by injection under the skin near the nipple. After you receive the injection, the radiologist will take more ultrasound images and videos of the tumor and lymph nodes in the underarm area.

You will have a biopsy of the sentinel lymph node that was identified in the ultrasound and a titanium clip marker will be inserted into the node. The clip helps distinguish the biopsied node from other nodes. You will be told the results of biopsy. After the biopsy, a radioactive seed may be inserted into the node to allow the surgeon to find and remove it during your surgery, an extra node may be removed at that time.

You will still have standard of care sentinel lymph node biopsy during your already scheduled surgery. You will sign a separate surgical consent form that explains this procedure and its risks.

You will be called by phone 30 days after the seed is removed to check for any side effects. This phone call should take about 10 minutes.

Length of Study:

Your active participation in this study will be over the follow up phone call.

This is an investigational study. Perflutren protein type A is FDA approved and commercially available for use in contrast-enhanced echocardiograms. Its use in this study is investigational.

Up to 21 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. Ipsilateral biopsy-proven invasive breast cancer <5 cm in maximal dimension by Ultrasound or Mammography.
3. No abnormal axillary nodes identified on grayscale AUS, or abnormal nodes with benign subsequent FNA biopsy.

Exclusion Criteria:

1. Pregnant or nursing women
2. Prior SLN dissection
3. Neoadjuvant chemotherapy.
4. Prior axillary lymph node surgery.
5. Prior history of ipsilateral breast cancer.
6. Known or suspected: Cardiac shunts
7. Known or suspected: hypersensitivity to perflutren, blood, blood products or albumin
8. Known or suspected: hypersensitivity to a prior OPTISON administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basak Dogan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 09, 2015 to February 22, 2016. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- CEUS SNL Imaging + Guided Biopsy: Subdermal periareolar injection of 0.2 - 0.5 cc of microbubble contrast Perflutren Protein-Type A Microspheres Injectable Suspension before Contrast-Enhanced Ultrasound (CEUS), sentinel lymph node (SNL) biopsy and radioactive seed placement.
Period: Overall Study
Arm/Group | CEUS SNL Imaging + Guided Biopsy
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- CEUS Sentinel Lymph Node Imaging + Guided Biopsy: Subdermal periareolar injection of 0.2 - 0.5 cc of microbubble contrast Perflutren Protein-Type A Microspheres Injectable Suspension before Contrast-Enhanced Ultrasound (CEUS), sentinel lymph node biopsy and radioactive seed placement.
Arm/Group | CEUS Sentinel Lymph Node Imaging + Guided Biopsy
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 62 [37 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Breast Cancer Participants With Sentinel Lymph Nodes (SLN) Identification Using the CEUS Technique
Description: Following the Microbubble CEUS of ipsilateral axillary nodes, needle biopsy and I-125 seed placement, a single node/participant (biopsied node) will be included in the statistical evaluation. The technique determined as technically feasible if an enhancing node is visualized in at least 90% of the subjects and 80% concordance is achieved between imaging-guided biopsy and final surgical histopathology. If no enhancement is identified, the overlying skin will be massaged, and re-injection of contrast will be employed up to three times. If no contrast enhancement in lymphatics is observed, the case will be reported as a failure of the CEUS technique.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | CEUS Sentinel Lymph Node Imaging + Guided Biopsy
Number analyzed (Participants) | 21
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the course of the CEUS SLN imaging and biopsy expected to all performed in a single interaction one day.
Arm/Group | CEUS Sentinel Lymph Node Imaging + Guided Biopsy
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEUS Sentinel Lymph Node Imaging + Guided Biopsy (N=21)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes